CLINICAL TRIAL: NCT01798329
Title: Minimal Hepatic Encephalopathy in Pre-hepatic Portal Hypertension Due to Portal Vein Thrombosis in Childhood and Young Adult: epidemiOlogical Study and Pilot Interventional Study.
Brief Title: ETOS: Minimal Hepatic Encephalopathy in Childhood and Young Adult: epidemiOlogical Study and Pilot Interventional Study
Acronym: ETOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Dr. Lorenzo D'Antiga, MD, Director of Pediatric Unit, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ETOS
Record Dates: First submitted 2013-02-19; First posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Hepatic Encephalopathy
Keywords: Minimal Hepatic Encephalopathy; Pre-hepatic Portal Hypertension; portal vein thrombosis
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Active Comparator): Probiotic VSL#3 for 15 weeks, dosage variations according to the weight
  Interventions: Dietary Supplement: probiotic VSL#3
- Placebo (Placebo Comparator): subjects treated with placebo for 15 weeks

INTERVENTIONS:
Dietary Supplement: probiotic VSL#3 — VSL#3 is a probiotic that reduces:
  * urease faecal activity
  * faecal pH
  * inflammatory cytokine
  Arms: Probiotic

SUMMARY:
The aim of the study is:

* Epidemiological/observational: investigating the presence of neuropsychological and electrophysiological alterations, suggesting a condition of minimal hepatic encephalopathy(and its behavioral correlates), in childhood and young adulthood affected by pre-hepatic portal hypertension due to portal vein thrombosis, even for implementing specific diagnostic protocols.
* Interventional: collecting preliminary data on the effects of a probiotic, in order to implement a controlled clinical study.

DETAILED DESCRIPTION:
Epidemiological/observational study investigating the presence of neuropsychological and electrophysiological alterations, suggesting a condition of minimal hepatic encephalopathy(and its behavioral correlates), in childhood and young adulthood affected by pre-hepatic portal hypertension due to portal vein thrombosis, even for implementing specific diagnostic protocols

ELIGIBILITY:
Inclusion Criteria:

* extra-hepatic portal vein thrombosis
* 4-20 years
* knowledge of italian language
* absence of perceptive or communicative deficit
* absence of psychiatric disease or mental retardation

Exclusion Criteria:

* medical contraindications for required evaluations
* infective pathologies
* parenchymal hepatic pathologies

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
neuropsychological and electrophysiological aspects | after 15 weeks of probiotic or placebo treatment
  Improvement in the spectrum of the digitalised electroencephalogram, improvement in the performance of the psychometric tests

SECONDARY OUTCOMES:
biochemical blood test | after 15 weeks of probiotic or placebo treatment
  Decreased level of serum ammonia
urine and faeces analysis | after 15 weeks of probiotic or placebo treatment
abdomen scan with color doppler technique | after 15 weeks of probiotic or placebo treatment
neurological evaluation | after 15 weeks of probiotic or placebo treatment
dietary anamnesis (last three days) | after 15 weeks of probiotic or placebo treatment
bowel frequency and characteristics | after 15 weeks of probiotic or placebo treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - University of Padua, Padua

REFERENCES:
- [Background] Amodio P, Montagnese S, Gatta A, Morgan MY. Characteristics of minimal hepatic encephalopathy. Metab Brain Dis. 2004 Dec;19(3-4):253-67. doi: 10.1023/b:mebr.0000043975.01841.de. PMID 15554421
- [Background] Amodio P, Campagna F, Olianas S, Iannizzi P, Mapelli D, Penzo M, Angeli P, Gatta A. Detection of minimal hepatic encephalopathy: normalization and optimization of the Psychometric Hepatic Encephalopathy Score. A neuropsychological and quantified EEG study. J Hepatol. 2008 Sep;49(3):346-53. doi: 10.1016/j.jhep.2008.04.022. Epub 2008 Jun 2. PMID 18602716
- [Background] Amodio P, Marchetti P, Del Piccolo F, de Tourtchaninoff M, Varghese P, Zuliani C, Campo G, Gatta A, Guerit JM. Spectral versus visual EEG analysis in mild hepatic encephalopathy. Clin Neurophysiol. 1999 Aug;110(8):1334-44. doi: 10.1016/s1388-2457(99)00076-0. PMID 10454268
- [Background] Amodio P, Del Piccolo F, Marchetti P, Angeli P, Iemmolo R, Caregaro L, Merkel C, Gerunda G, Gatta A. Clinical features and survivial of cirrhotic patients with subclinical cognitive alterations detected by the number connection test and computerized psychometric tests. Hepatology. 1999 Jun;29(6):1662-7. doi: 10.1002/hep.510290619. PMID 10347105